CLINICAL TRIAL: NCT01307787
Title: Effects of a Group-based Exercise and Educational Program on Physical Performance and Disease Self-management in Rheumatoid Arthritis: a Randomized Controlled Study
Brief Title: Effects of a Rehabilitation Program on Physical Performance and Disease Self-management in Rheumatoid Arthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: E.van Weert, UMCG
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 210.076
Record Dates: First submitted 2011-03-02; First posted 2011-03-03 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Rheumatoid Arthritis
Keywords: exercise; education; self-management; rehabilitation
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fit-program (Experimental): Participants in the intervention group followed an eight week multi-disciplinary group rehabilitation program, consisting of a physical exercise part and an educational component.
  Interventions: Other: experimental Fit-program
- waiting list control group (Other): The waiting-list control group was allowed to enter the FIT program for rehabilitation after the study period.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: experimental Fit-program — Participants in the intervention group followed an eight week multi-disciplinary group rehabilitation program, consisting of a physical exercise part and an educational component. The physical exercise part consisted of a muscle exercise circuit and bicycle training,sport and aqua jogging. The educational part consisted of a weekly sixty minutes session. A multi-disciplinary group of healthcare professionals gave specialist orientated informational advice about how to handle the consequences of RA. Special attention was paid to ensure adjusting the level of each patients activity level to the participants' actual energy level. Further information was given about body sensations, sports, food and energy, pain, fatigue, emotional changes, sleeping disturbance and daily routine.
  Other Names: rehabilitation
  Arms: fit-program
Other: no intervention — waiting list control group with no intervention
  Other Names: rehabilitation
  Arms: waiting list control group

SUMMARY:
The purpose of this study is to evaluate the effects of a group-based exercise and educational program for people with Rheumatoid Arthritis (RA) on physical performance and disease-self-management.

DETAILED DESCRIPTION:
Currently, the effectiveness of a program consisting of education to improve disease self-management combined with intensive exercises is not clear. In the present study the investigators developed a group-based program for people with RA consisting of physical exercise to increase physical performance (i.e. aerobic capacity and muscle strength) combined with an educational program to improve disease self-management (self-reported health status and self-efficacy). The investigators called it the 'FIT program'. The aim of the present randomized controlled trial (RCT) was to examine the effects of the FIT program on aerobic capacity, muscle strength, self-reported health status and self-efficacy, in a population of people with RA. The investigators hypothesized that the FIT-program would have beneficial effects on physical performance (ie. aerobic capacity and muscle strength) and disease self-management (i.e. perceived health status and self-efficacy components) compared to a waiting list control group (WLCgroup).

ELIGIBILITY:
Inclusion Criteria:

* medical diagnosis of RA according to the American College of Rheumatology (ACR) criteria
* between 18 and 66 years of age

Exclusion Criteria:

* severe disease activity (Disease Activity Score:DAS-28 > 5.1)
* cardiac or pulmonary diseases resulting in restrictions in their ability to follow a physical exercise program
* a Steinbrocker classification of functional capacity in RA ≥ 3
* no stable medication for the RA
* intra-articular injections during the time of the study

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen van Weert, phd, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Center for Rehabilitation, Haren, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Breedland I, van Scheppingen C, Leijsma M, Verheij-Jansen NP, van Weert E. Effects of a group-based exercise and educational program on physical performance and disease self-management in rheumatoid arthritis: a randomized controlled study. Phys Ther. 2011 Jun;91(6):879-93. doi: 10.2522/ptj.20090010. Epub 2011 Apr 7. PMID 21474637

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Rheumatologist referred people diagnosed with RA to the rehabilitation department if they had complaints concerning their physical performance or if they experienced problems with the daily management of their illness. Referred participants were independent and living at home. They did not include residents of nursing homes.
Pre-assignment Details: A total of thirty-nine individuals were referred for this study. Thirty-four individuals returned a signed Informed Consent form and five decided not to participate for a variety of reasons.(Impairment due to trauma n = 1 Not able to follow the program n = 1 Personal reasons n = 3)
Groups:
- Fit-program: Participants in the intervention group followed an eight week multi-disciplinary group rehabilitation program, consisting of a physical exercise part and an educational component. The physical exercise part took place in group sessions and consisted of a muscle exercise circuit and bicycle training once a week for sixty minutes, sport once a week for sixty minutes and aqua jogging twice a week for thirty minutes.
  The educational part consisted of a weekly sixty minutes session. A multi-disciplinary group of healthcare professionals consisting of a psychologist, physical therapist, occupational therapist, dietician and a social worker gave specialist orientated informational advice about how to handle the consequences of RA. Special attention was paid to ensure adjusting the level of each patients activity level to the participants' actual energy level.
- Waiting List Control Group: The waiting list control group did not have an intervention during the evaluation part of the study.The waiting-list control group was allowed to enter the FIT program for rehabilitation after the study period.
Period: Overall Study
Arm/Group | Fit-program | Waiting List Control Group
Started | 19 | 15
T1= After 9 Weeks Post Intervention | 18 | 15
T2= After 22 Weeks at Follow-up | 17 | 15
Completed | 17 | 15
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fit-program | Waiting List Control Group | Total
Number analyzed (Participants) | 19 | 15 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 15 | 34
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (11.9) | 51.8 (9.4) | 48 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 7 | 3 | 10
Region of Enrollment [Number; unit: participants]
  Netherlands | 19 | 15 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in VO2 Max, Maximum Oxygen Uptake in ml/Min/kg is the Standard Index of Cardio-respiratory Fitness
Description: maximum oxygen uptake(VO2max, in ml/min/kg)was determined using the Åstrand-Rhyming test.The workload on the cycle ergometer was increased every minute by 25 watts until a steady-state heart rate was achieved. Participants had to sustain cycling for about 6 minutes, the heart rate(HR) was taken every minute. Mean HR of the 5th and 6th minute was registered. With the given workload, observed HR and participants'weight, maximal oxygen uptake can be established using the Åstrand-Rhyming nomogram. Values vary from < 21( sedentary with disease) to > 57 ( very good physical condition).
Time Frame: baseline, postintervention at 9 weeks
Population: Some VO2 max data (n=4 in the intervention group and n=2 in the WLC group)could not be collected because of specific participant conditions at different testing time points. 4 subjects did not reach the necessary heart rate to estimate the VO2 max. One subject had hypertension and one subject had knee problems.
Measure: Mean (Standard Deviation); unit: ml/min/kg
Groups:
- Intervention Fit Program: An eight week multi-disciplinary group-therapy program for people with RA, consisting of physical exercise designed to increase aerobic capacity and muscle strength together with an educational program to improve health status and self-efficacy for disease-self-management.
- Waiting List Control Group: No intervention. The waiting-list control group was allowed to enter the FIT program for rehabilitation after the study period.
Arm/Group | Intervention Fit Program | Waiting List Control Group
Number analyzed (Participants) | 15 | 13
ml/min/kg | 3.82 (3.86) | -0.44 (2.21)
Statistical Analysis 1: Comparison: Intervention Fit Program vs Waiting List Control Group; Mann-Whitney U tests were used to assess between group changes on delta scores at times T0( at the start of the study in week 1) and T1( post-intervention in week 9). Significance level for all statistical tests was set at p< 0.05; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Self-efficacy Pain and Other Symptoms
Description: Self-efficacy was assessed by the Arthritis-Self-efficacy Scale Dutch version. This arthritis self-efficacy scale contains two sub scales: self-efficacy pain (5 items related to coping with pain, and self-efficacy other symptoms (6 items related to coping with other symptoms, such as depression, fatigue and frustrations.A five-point ordinal scale is used ranging from 'totally disagree' (1) to 'totally agree' (5). We computed a mean score of 11 items ranging from 1-5. A higher score refers to higher self-efficacy.
Time Frame: baseline, postintervention at 9 weeks,
Population: per protocol 2 subjects( n=2) in the intervention fitprogram withdrew from the study
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention Fit Program: Participants in the intervention group followed an eight week multi-disciplinary group rehabilitation program, consisting of a physical exercise part and an educational component.
- Waiting List Control Group: no intervention. WLC was allowed to follow the program after the study.
Arm/Group | Intervention Fit Program | Waiting List Control Group
Number analyzed (Participants) | 17 | 15
units on a scale | 0.42 (0.71) | 0.28 (0.85)
Statistical Analysis 1: Comparison: Intervention Fit Program vs Waiting List Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.47, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Self-efficacy Function
Description: Self-efficacy function was assessed by the Arthritis-Self-efficacy Scale Dutch version The subscale self-efficacy function contains 8 items related to physical function. A five-point ordinal scale is used ranging from 'totally disagree' (1) to 'totally agree' (5). A mean score of 8 items was computed ranging from 1-5. A higher score refers to higher self-efficacy.
Time Frame: baseline, postintervention at 9 weeks,
Population: analysis per protocol, 2 subjects(n=2) in the intervention fitprogram withdrew from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention Fitprogram Group: Participants in the intervention group followed an eight week multi-disciplinary group rehabilitation program, consisting of a physical exercise part and an educational component.
- Waiting List Control Group: no intervention, allowed to follow the program after the study
Arm/Group | Intervention Fitprogram Group | Waiting List Control Group
Number analyzed (Participants) | 17 | 15
units on a scale | 0.29 (0.57) | 0.10 (0.38)
Statistical Analysis 1: Comparison: Intervention Fitprogram Group vs Waiting List Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.24, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Muscle Strength of the Upper Extremity
Description: Muscle strength was assessed using a hand-held dynamometer (Microfet, Hoggan health Industries Inc.USA).Maximal voluntary isometric muscle strength of the elbow-flexors, elbow-extensors, was tested and recorded three times for each muscle group. All tests were performed bilaterally. The mean value of three measurements was computed. In addition a sum score of the mean values of the flexors and extensors on both sides for the upper extremity (UE)was computed and taken for analyses.
Time Frame: baseline, postintervention at 9 weeks,
Population: per protocol, one subject (n=1) in the intervention fitprogram withdrew from the study.
Measure: Mean (Standard Deviation); unit: newton
Arm/Group | Intervention Fitprogram Group | Waiting List Control Group
Number analyzed (Participants) | 18 | 15
newton | 36.06 (121.71) | -5.49 (96.46)
Statistical Analysis 1: Comparison: Intervention Fitprogram Group vs Waiting List Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.16, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Muscle Strength of the Lower Extremity
Description: Muscle strength was assessed using a hand-held dynamometer (Microfet, Hoggan health Industries Inc.USA).Maximal voluntary isometric muscle strength of the knee-flexor and knee-extensors, was tested and recorded three times for each muscle group. All tests were performed bilaterally. The mean value of three measurements was computed. In addition a sum score of the mean values of the flexors and extensors on both sides for the lower extremity (LE)was computed and taken for analyses.
Time Frame: baseline, postintervention at 9 weeks,
Population: per protocol,Lower extremity(LE) muscle strength data for one participant(n=1) in the WLC group is missing because knee problems prevented testing.
Measure: Mean (Standard Deviation); unit: newton
Arm/Group | Intervention Fitprogram Group | Waiting List Control Group
Number analyzed (Participants) | 18 | 14
newton | 111.20 (184.82) | 25.61 (189.30)
Statistical Analysis 1: Comparison: Intervention Fitprogram Group vs Waiting List Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.21, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Health Status: Physical Health
Description: Self-reported health status was assessed using the Arthritis Impact-Measurement Scale-2, the Dutch version (Dutch-AIMS2).The questionnaire contains 77 items which represent 5 dimensions: physical functioning, psychological functioning, symptoms, social interaction and role functioning. Responses are recorded on a 5-point scale. All responses were recoded and calculated to a 0-10 scale. Scores were modified according to the number of co-morbidity complaints, as was recommended in the Dutch-AIMS2 manual. A low score indicates better health.
Time Frame: baseline, postintervention at 9 weeks,
Population: per protocol,2 subjects( n=2) in the intervention fitprogram withdrew from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Fitprogram Group | Waiting List Control Group
Number analyzed (Participants) | 17 | 15
units on a scale | -0.68 (1.00) | -0.14 (0.49)
Statistical Analysis 1: Comparison: Intervention Fitprogram Group vs Waiting List Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.07, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in Health Status: Psychological Health
Description: as for outcome 6
Time Frame: baseline, postintervention at 9 weeks,
Population: analysis per protocol,2 subjects( n=2) in the intervention fitprogram withdrew from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Fitprogram Group | Waiting List Control Group
Number analyzed (Participants) | 17 | 15
units on a scale | -0.34 (1.11) | 0.08 (1.37)
Statistical Analysis 1: Comparison: Intervention Fitprogram Group vs Waiting List Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Change in Health Status: Social Interaction
Description: as for outcome 6
Time Frame: baseline, postintervention at 9 weeks,
Population: per protocol,2 subjects( n=2) in the intervention fitprogram withdrew from the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Fitprogram Group | Waiting List Control Group
Number analyzed (Participants) | 17 | 15
units on a scale | -0.48 (1.90) | -0.88 (2.03)
Statistical Analysis 1: Comparison: Intervention Fitprogram Group vs Waiting List Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Description: serious and other non-serious adverse events were not collected/assessed.
Arm/Group | Fit-program | Waiting List Control Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
An important limitation in our study was the low number of participants included in both groups which may have induced a lack of power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes